CLINICAL TRIAL: NCT00086840
Title: A Phase II Study of CCI-779 in Patients With Relapsed, Refractory or Transformed Chronic Lymphocytic Leukemia
Brief Title: CCI-779 in Treating Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02598; MDA-2003-0886; N01CM17003 (NIH); CDR0000371619 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — temsirolimus; Sirolimus

ARMS (1):
- Treatment (temsirolimus) (Experimental): Patients receive CCI-779 IV over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving an objective response may receive 3 consolidation courses of therapy.
  Interventions: Drug: temsirolimus; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well CCI-779 works in treating patients with relapsed or refractory chronic lymphocytic leukemia. Drugs used in chemotherapy, such as CCI-779, work in different ways to stop cancer cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the activity of CCI-779 in patients with relapsed, refractory, or transformed chronic lymphocytic leukemia.

OUTLINE: Patients are stratified according to disease (relapsed or refractory chronic lymphocytic leukemia [CLL] vs transformed CLL).

Patients receive CCI-779 IV over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving an objective response may receive 3 consolidation courses of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic lymphocytic leukemia (CLL)

  * Relapsed, refractory, or transformed disease

    * Relapsed disease defined as symptomatic loss of a prior partial or complete response to a regimen containing a purine analog and/or a monoclonal antibody AND evidence of disease progression
    * Primary resistant disease defined as failure to achieve an objective response to a regimen containing a purine analog and/or a monoclonal antibody
    * Transformed CLL (Richters transformation), must meet both of the following criteria:

      * Histologically confirmed lymphoma
      * Measurable disease
* No CNS disease
* Performance status - ECOG 0-2
* Bilirubin ≤ 2 mg/dL (unless elevated due to Gilbert's disease)
* SGOT and SGPT < 3 times upper limit of normal
* Creatinine ≤ 2 mg/dL (unless due to organ leukemic involvement)
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV-positive patients allowed provide CD4 counts are normal and no AIDS-defining disease is present
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to CCI-779
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent uncontrolled illness
* See Disease Characteristics
* No concurrent prophylactic hematopoietic colony-stimulating factors
* See Disease Characteristics
* More than 2 weeks since prior cytotoxic chemotherapy and recovered
* More than 2 weeks since prior radiotherapy and recovered
* No other concurrent investigational or antitumor agents
* No other concurrent cytotoxic agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-05; Primary Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Response (CR or PR) | 6 months
  Defined as the complete disappearance of all known disease, or a 50% decrease in tumor size using the sum of the product (bi-perpendicular dimensions when available).

CONTACTS AND LOCATIONS:
Overall Officials: Francis Giles, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States